CLINICAL TRIAL: NCT06673719
Title: Comparative Validity of 99mTc-pertechnetate SPECT/CT and Mean Intragastric Pressure During Nutrient Drink in the Measurement of Gastric Accommodation
Brief Title: Comparing Pertechnetate SPECT/CT and Intragastric Pressure During Nutrient Drink for Gastric Accommodation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Nashrulhaq Tagiling, MSc, Principal Investigator, Universiti Sains Malaysia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: USM/JEPeM/19040249
Record Dates: First submitted 2024-10-30; First posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-10

CONDITIONS: Healthy Volunteers; Functional Dyspepsia

STUDY DESIGN:
Intervention Model Description: Monocentric, non-randomized sequence, pilot and feasibility study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- SPECT/CT or HRM-NDT (Experimental)
  Interventions: Radiation: 99mTc-pertechnetate SPECT/CT; Procedure: Combined High-Resolution Manometry-Nutrient Drink Test

INTERVENTIONS:
Radiation: 99mTc-pertechnetate SPECT/CT — This procedure is similar to standard Meckel's diverticulum scan, with the addition of SPECT/CT acquisition to measure gastric volume.
Procedure: Combined High-Resolution Manometry-Nutrient Drink Test — Proximal gastric high-resolution manometry was done concurrently with nutrient drink test to measure proximal gastric function.

SUMMARY:
Functional dyspepsia (FD) is a common gastrointestinal disorder which can present with early satiety, postprandial fullness, epigastric pain and burning sensation in the absence of underlying disease. The most troubling symptom is weight loss, prevalent in up to 40% of FD patients and is often associated with impaired gastric accommodation.

Gastric accommodation by definition is a reflex, mediated vagally which causes reduction in gastric tone, increased in compliance and increment in gastric volume post meal ingestion. It allows large volumes of liquid or solid ingestion without causing postprandial symptoms. Impairment of gastric accommodation has been linked to gastrointestinal symptoms which includes nausea, bloating, early satiety, weight loss and epigastric pain.

There are several studies aimed to assess efficacy in the treatment of functional dyspeptic patients. A myriad of tests can measure gastric accommodation such as gastric barostat and single photon emission computed tomography (SPECT). An alternative study known as the nutrient drink test has also been proposed and can be combined with high-resolution manometry.

So far, none of the nuclear medicine centers in Malaysia are providing clinical service for radionuclide gastric accommodation study. The gold standard for gastric accommodation assessment is the gastric barostat method. However, the technique is invasive and caused discomfort to patients. Radionuclide gastric accommodation study using 99mTc-pertechnetate with SPECT/CT is a non-invasive method that can be used to assess patient with FD and enables quantitative evaluation of treatment response to medications. Hence, the role of non-invasive gastric volume assessment with 99mTc-pertechenate SPECT/CT in the evaluation of healthy individuals was studied first, and then compared with intragastric pressure measurements from high-resolution manometry and nutrient drink test.

ELIGIBILITY:
Healthy volunteers

Inclusion Criteria:

* Patient is above 18 years-old.
* No current gastrointestinal symptoms
* No previous gastrointestinal illness such as peptic ulcer disease or gastritis
* No chronic medical illness such as chronic neurological, cardiovascular, pulmonary, endocrine and hematological disorders
* Does not fulfill Rome IV criteria for functional dyspepsia

Exclusion Criteria:

* • Had undergone any abdominal surgery except appendicectomy, tubal ligation or Caesarean section

  * Use of medications such as metoclopramide, domperidone, erythromycin and itopride that may alter gastrointestinal function and motility
  * Pregnant woman

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-02-27 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
Number of participants completing each procedure | From the initiation of the first study procedure until the completion of the second procedures (up to 30 days)
  • Feasibility assessed as technical success (number of participants completing each procedure).
Duration (time) of each procedural session | From the initiation of the first study procedure until the completion of the second procedures (up to 30 days)
  • Feasibility assessed as procedural duration (time taken to complete one procedure)
Incidence of adverse event | From the initiation of the first study procedure until the completion of the second procedures (up to 30 days)
  • Tolerability assessed as incidence of adverse event over study period using the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

SECONDARY OUTCOMES:
Gastric volume measured using SPECT/CT | During the procedure, 1 day
  • Gastric volume (in mL): Fasting state, postprandial state (after single-serving of 250 mL nutrient drink). All are to be measured in one session and as one outcome.
Proximal gastric pressure measured using high-resolution manometry | During the procedure, 1 day
  • Proximal gastric pressure (in mmHg): baseline (fasting) pressure recording, prandial pressure recording, postprandial pressure recording. All are to be measured in one session and as one outcome.
Nutrient drink tolerance | During the procedure, 1 day
  • Maximum tolerated volume (in mL): Number of drink volume required to achieve satiety
Dyspeptic symptoms measured using numerical rating scales | During the procedure, 1 day
  • Dyspeptic symptom responses: Numerical rating scale with verbal descriptors on 4 symptoms i.e., epigastric pain, bloating, fullness, nausea (from 0 to 3: 0 means "no symptoms", 3 means "severe"). All are to be measured in one session using one instrument and as one outcome.
Satiation score measured using numerical rating scales | During the procedure, 1 day
  • Satiation (presented as satiation-unit): Numerical rating scale with verbal descriptors (from 0 to 5: 0 means "not full", 5 means "maximum fullness")

CONTACTS AND LOCATIONS:
Overall Officials: Yeong Yeh Lee, MD, PhD, Study Director — Universiti Sains Malaysia
Locations (1):
- Universiti Sains Malaysia, Kota Bharu, Kelantan, Malaysia

IPD SHARING:
Plan to Share IPD: Undecided